CLINICAL TRIAL: NCT07195253
Title: Exploring the Relationships Between Oro-myofunctional Characteristics and Obstructive Sleep Apnea in Infants With Down Syndrome
Brief Title: Oro-myofunctional Characteristics and Obstructive Sleep Apnea in Infants With Down Syndrome
Acronym: OMF21
Status: Not yet recruiting | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL25_0309; 2025-A01900-49 (Other: ID-RCB)
Record Dates: First submitted 2025-09-02; First posted 2025-09-26 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Obstructive Sleep Apnea; Down Syndrome (Trisomy 21)
Keywords: sleep apnea; Down Syndrome; oro-myofunctional development; sleep; non-nutritive sucking
MeSH Terms: conditions — Sleep Apnea, Obstructive; Down Syndrome; Sleep Apnea Syndromes | interventions — Polysomnography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Infants with Down Syndrome: 6 month-old infants with Down Syndrome recorded by polysomnography
  Interventions: Diagnostic Test: Polysomnography (PSG) to explore OSA; Other: Oro-myo-functional clinical evaluation; Other: Sleep Disturbance Scale for Children; Other: Non-nutritive sucking recording; Behavioral: Neurocognitive evaluation; Other: PedsQL-Infants; Other: Sleep Hygiene Scale for Children

INTERVENTIONS:
Diagnostic Test: Polysomnography (PSG) to explore OSA — Patients will undergo full-night PSG (including electrocardiogram to monitor heart rate and the JAWAC system to record mandibular movements) in the sleep unit of Hôpital Femme-Mère-Enfant (Bron, France) to explore OSA, included in the routine care of children with DS.
  OSA diagnosis will be made based on the obstructive apnea-hypopnea index (OAHI) resulting from the PSG. OSA will be diagnosed when OAHI ≥1.5/hour.
Other: Oro-myo-functional clinical evaluation — Orofacial myofunctional evaluation will be conducted by a physiotherapist according to the OMES-E (Orofacial Myofunctional Evaluation with Scores for Nursing Infants).
Other: Sleep Disturbance Scale for Children — The Sleep Disturbance Scale for Children is a short questionnaire answered by parents about their child's sleep disorders.
  Total score and scores for each sleep disorder will be calculated, according to the classical procedures during hospitalization of all children in our sleep unit.
Other: Non-nutritive sucking recording — Non-nutritive sucking performance will be recorded through an experimental method using a classical pacifier, equipped with pressure sensors. Recording will last about 10 minutes. Variables related to sucking performance (maximum amplitude, frequency of sucking bursts, etc.) will be recorded.
Behavioral: Neurocognitive evaluation — The Bayley Scales of Infant and Toddler Development (4th edition) will be administered by a neuropsychologist. Five subset scores (cognitive, receptive communication, expressive communication, fine motor, gross motor) will be calculated, along with three composite scores (cognitive, language, motor).
Other: PedsQL-Infants — The PedsQL-Infants questionnaire is designed to evaluate quality of life in infants. It will be given to parents during their child's hospitalization.
Other: Sleep Hygiene Scale for Children — The Sleep Hygiene Scale for Children is a short questionnaire answered by parents about behavioral sleep disorders.
  Total result ("sleep hygiene issue" : yes/no) and three scores (attachment parenting, translational coping, screen exposure) will be calculated, according to the classical procedures during hospitalization of all young children in our sleep unit.

SUMMARY:
Obstructive Sleep Apnea (OSA) is characterised by repetitive collapse of the upper airway during sleep, inducing breathing disturbances that can result in oxygen desaturation and frequent arousals. In children, OSA can have long-term consequences on the development and on the cardiovascular system.

Down Syndrome (DS) is a genetic disorder associated with intellectual disability and many comorbidities. The prevalence of OSA is particularly high in patients with DS, from infancy. In a recent study by Fauroux et al. (2024), OSA was diagnosed in 97% infants and early diagnosis and intervention from the age of 6 months was associated with better neurocognitive outcome at 3 years old. However, polysomnography (PSG - the gold standard method for diagnosing OSA) is poorly accessible, highlighting the need to develop new strategies to prevent and to screen OSA early in infancy.

OSA can be linked to some orofacial abnormalities presented by patients with DS. Indeed, orofacial functions and structures ca play a crucial role in OSA. For example, nose breathing allows the tongue to act as a stimulator of the transverse maxillary growth during childhood, allowing the upper airway to develop properly.

The primary objective of the present study is to explore the relationships between oro-myo-facial functions, more specifically non-nutritive sucking, and the severity of OSA in 6 months old infants with DS.

The main hypothesis is that OSA severity (estimated by the obstructive apnea hypopnea index on PSG) will be negatively correlated to non-nutritive sucking performance.

Data from this study could help developing easily accessible protocols for OSA screening based on simple sucking recording. Some interventions could also be tested to prevent OSA from the beginning of life, like an innovative pacifier recently developed by a French start-up to stimulate nose breathing and to promote correct positioning of the tongue.

ELIGIBILITY:
Inclusion Criteria:

(infants with Down Syndrome)

* Aged 6 months (±3 weeks)
* Diagnosed with Trisomy 21
* Affiliated to a social security scheme
* With informed consent of the 2 legal representatives

Exclusion Criteria:

* Diagnosed with mosaic Down syndrome
* Born preterm (gestation age at birth <37 weeks)
* Treated for OSA with Continuous Positive Airway Pressure
* Known allergy to silicone
* Currently participating to an interventional study protocol implying an ongoing exclusion period from other studies
* Refusal from legal representatives.

Ages: 5 Months to 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: This study involves 6-month-old infants diagnosed with Down syndrome.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2027-10 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Number of peaks composing sucking bursts and obstructive apnea-hypopnea index (OAHI) | Day 1
  Number of peaks during sucking bursts will be measured by non-nutritive sucking recording.
  OAHI will be measured by PSG.

SECONDARY OUTCOMES:
Oro-facial myo-functional characteristics | D1
  Variables obtained from electrophysiological (non-nutritive sucking recording) and clinical (OMES-E: 1 total score + 12 subscores) examination of oro-facial myo-functional characteristics.
Respiratory PSG indices | Night between Day 1 and Day 2.
  Obstructive apnea-hypopnea index (OAHI), apnea-hypopnea index (AHI), respiratory effort-related arousal index (RERA), mean CO2, time spent with CO2 >50mmHg, mean SpO2, desaturation index >3%, pulse wave amplitude drop (PWAD), hypoxic burden.
  PSG sleep architecture parameters: total sleep time (TST), sleep efficiency (TST / time in bed), sleep onset latency (SOL), wake after sleep onset (WASO), percentage of sleep stages (N1, N2, N3, REM), arousal index, awakening index, mandibular movement index.
Subjective parental evaluation of sleep disorders on the Sleep Disturbance Scale for Children (SDSC) | Day 1
  SDSC: 1 total score and subscores (insomnia, sleep disordered breathing, non-restorative sleep)
Subjective parental evaluation of sleep hygiene on the Sleep Hygiene Scale for Children (SHSC) | Day 1
  1 total result ("sleep hygiene issue" : yes/no) and three scores (attachment parenting, translational coping, screen exposure)
Heart rate variability (HRV) | Night between Day 1 and Day 2.
  Time-domain HRV indices: RR, HR, NN50, pNN50, SDNN, RMSSD Frequency-domain HRV indices: Ptot, VLF, LF, HF, LFnu, HFnu, LF/HF ratio. HRV measures will be compared between the sample of children with DS and a control group of healthy children from the AuBE cohort.
Electrophysiological evaluation of sucking | Day 1
  All other variables obtained from non-nutritive sucking recording
Neuropsychological evaluation | Day 2
  Neurosychological evaluation will be conducted by an experienced neuropsychologist using the Bayley Scales of Infant and Toddler Development (4th edition). Total score and subscores (posture, hand-eye coordination, language, sociability) will be collected.
Quality of life on the PedsQL | Day 1
  Results of the PedsQL consist in 1 total score + 5 subscores (physical functioning, physical symptoms, emotional functioning, social functioning, cognitive functioning)
Clinical examination of oro-facial myo-functional characteristics | Day 2
  Variables obtained from clinical examination of oro-facial myo-functional characteristics driven by an experienced physiotherapist following the Expanded protocole of Orofacial Myofunctional Evaluation with Scores (OMES-E).
PSG sleep architecture parameters | Night between Day 1 and Day 2.
  Total sleep time (TST), sleep efficiency (TST / time in bed), sleep onset latency (SOL), wake after sleep onset (WASO), percentage of sleep stages (N1, N2, N3, REM), arousal index, awakening index, mandibular movement index

CONTACTS AND LOCATIONS:
Locations (1):
- Service d'épileptologie clinique, des troubles du sommeil et de neurologie fonctionnelle de l'enfant, Bron, France